CLINICAL TRIAL: NCT06202963
Title: Has Ultrasound-guided Hydrorelease of Coracohumeral Ligamet Additional Benefit in Patients With Adhesive Capsulitis Receiving Ultrasound-guided Shoulder Hyrodilatation?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haydarpasa Numune Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sibel süzen Özbayrak, M.D., Haydarpasa Numune Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HNEAH-KAEK/KK/2023/210
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Adhesive Capsulitis
Keywords: Adhesive Capsulitis, Coracohumeral ligament, Hydrorelease, Hydrodilatation
MeSH Terms: conditions — Bursitis | interventions — Triamcinolone Acetonide; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): In group 1, hydrodilatation will be performed with intra-articular 40 mg triamcinolone, lidocaine, and physiological saline through a posterior approach to the shoulder, guided by ultrasonographic imaging. Fluid injection will continue until distension is observed in the shoulder joint capsule by ultrasonography. The amount of fluid given will be recorded.
  Interventions: Drug: Triamcinolone Acetonide
- Group 2 (Active Comparator): The second group will undergo hydrodilatation with intra-articular 40 mg triamcinolone, lidocaine, and physiological saline through a posterior approach to the shoulder, guided by ultrasonographic imaging. The amount of fluid given will be recorded. Additionally, with ultrasonographic evaluation, 2 cc of physiological saline will be injected into the corocohumeral ligament.
  Interventions: Drug: Triamcinolone Acetonide

INTERVENTIONS:
Drug: Triamcinolone Acetonide — 1. group will receive ultrasound-guided hydrodilatation
  2. group will receive ultarsound-guided coracohumeral hydrorelease in addition to the ultrasound-guided hydrodilaltation of shoulder
  Other Names: lidocaine; serum physiologic

SUMMARY:
The goal of this study is to detect if there is an additional benefit to performing ultrasound-guided hydrorelease of the coracohumeral ligament in patients with adhesive capsulitis of the shoulder receiving ultrasound-guided hydrodilatation.

DETAILED DESCRIPTION:
This study is organised as double-blind, randomised controlled trial. Written informed consent will be taken from all the patients participating to the study.

Inclusion Criteria

Patients between the ages of 30 and 70, who have complaints of shoulder pain and limitation in the shoulder for at least 3 months and are diagnosed with Adhesive Capsulitis by clinical examination, will be included in the study.

Exlusion Criteria

1. A history of physical therapy or injections for the shoulder joint within the previous three months,
2. The existence of a neurological condition or surgical history that could impair upper limb functions,
3. Being a breastfeeding or pregnant woman,
4. Mental illnesses and cognitive impairments that impair cooperation
5. Diabetes mellitus with unregulated glucose levels
6. Presenece of Cancer

Patients included in the study will be divided into two groups by block randomization.

In group 1, hydrodilatation will be performed with intra-articular 40 mg triamcinolone, lidocaine, and physiological saline through a posterior approach to the shoulder, guided by ultrasonographic imaging. Fluid injection will continue until distension is observed in the shoulder joint capsule by ultrasonography. The amount of fluid given will be recorded.

The second group will undergo hydrodilatation with intra-articular 40 mg triamcinolone, lidocaine, and physiological saline through a posterior approach to the shoulder, guided by ultrasonographic imaging. Additionally, with ultrasonographic evaluation, 2 cc of physiological saline will be injected into the corocohumeral ligament.

All the patients will be evaluated by a doctor who is blind to the study groups. Demographic information, history of shoulder pain, presence of chronic diseases, pain severity measured by VAS during resting,activity and sleep will be recorded. Physical examination including shoulder range of motion, will be evaluated. Shoulder Disability Index will be used for evaluating the functional status of shoulder. They will be evaluated before and immediately after injection, 1 week later, 1 month and 3 months after injection with VAS, shoulder range of motion and Shoulder Disability Index.

ELIGIBILITY:
Inclusion Criteria:

Patients between the ages of 30 and 70 who have complained of shoulder pain and limitation in the shoulder for at least 3 months and have been diagnosed with adhesive capsulitis by clinical examination will be included in the study.

Exclusion Criteria:

1. A history of physical therapy or injections for the shoulder joint within the previous three months,
2. The existence of a neurological condition or surgical history that could impair upper limb functions,
3. Being a breastfeeding or pregnant woman,
4. Mental illnesses and cognitive impairments that impair cooperation
5. Diabetes mellitus with unregulated glucose levels
6. Presence of Cancer

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Visual Analouge Scale (VAS) | Before and immediately after injection, 1 week,1 month and 2 moths after injection
  Pain Severity
Shoulder Range of Motion | Before and immediately after injection, 1 week,1 month and 2 moths after injection
  Shoulder Limitation
Shoulder Disability Index | Before injection, 1 week,1 month and 2 moths after injection
  Shouler Disability

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University Haydarpasa Numune Research and Training Hospital, Istanbul, Uskudar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided